CLINICAL TRIAL: NCT06471049
Title: Prospective, Controlled, Randomized Study Evaluating the Success Rate of Outpatient Management of the Total Benign Hysterectomy by Transvaginal Natural Orifice Transluminal Endoscopic Surgery (vNOTES) Compared to Each of the Two Laparoscopic Routes (Conventional and Robot-assisted).
Brief Title: Study Evaluating the Success Rate of Outpatient Management of the Total Benign Hysterectomy by Transvaginal Natural Orifice Transluminal Endoscopic Surgery (vNOTES) Compared to Each of the Two Laparoscopic Routes (Conventional and Robot-assisted).
Acronym: HYSTERAMBU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A02112-43
Record Dates: First submitted 2024-06-12; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Surgery; Gynecologic Disease
Keywords: hysterectomy; vnotes; laparoscopy
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transvaginal Natural Orifice Transluminal Endoscopic Surgery (vNOTES) (Experimental)
  Interventions: Procedure: Benign Hysterectomy
- Conventional laparoscopy (Active Comparator)
  Interventions: Procedure: Benign Hysterectomy
- Robot-assisted laparoscopy (Active Comparator)
  Interventions: Procedure: Benign Hysterectomy

INTERVENTIONS:
Procedure: Benign Hysterectomy — removal of the uterus

SUMMARY:
Benign total hysterectomy is one of the most commonly performed gynecological surgery.

Conventionally performed by a classical surgical approach, it is now provided routinely and for several years by laparoscopy and more recently by Robotic-Assisted Laparoscopy.

A third minimally invasive option is currently being developed and proposed to avoid trans-peritoneal access, using a vaginal trans-laparoscopic technique, defined by the name V-NOTES (Vaginal-Natural Orifice Transluminal Endoscopic Surgery).

These minimally invasive approaches have simplified this intervention on many surgical and anesthetic parameters (signing, surgical trauma, pain and post-operative ileus, recovery of autonomy) and consider possible management in the outpatient sector.

This study aims at enrolling women for which a total hysterectomy with or without annexectomy for the treatment of a benign pathology must be scheduled.

The objective of the study is to compare the success rate of outpatient treatment of the V-Notes route and the conventional laparoscopic route and to compare the success rate of outpatient treatment of the V-Notes route and the laparoscopic route assisted robot.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged 18 years old and over
* Participant for whom a total hysterectomy with or without adnexectomy for the treatment of a benign pathology must be scheduled
* Participant with no contraindication to being operated on by one of the three approaches under study (conventional laparoscopy, V-Notes, robot-assisted laparoscopy)
* Patient eligible for outpatient treatment
* Participant affiliated or beneficiary of a social security regimen
* Participant having been informed and having given her free, informed and written consent (at the latest on the day of inclusion and before any examination required by the research)

Exclusion Criteria:

* Participant with endometriosis with procedure associated with hysterectomy (digestive procedure, extended adhesiolysis, or other procedure)
* Participant whose physical and/or psychological health is severely impaired, which according to the investigator may affect the participant's understanding and compliance with the study
* Participant in another research
* Participant in a period of exclusion from another research still in progress at the time of inclusion
* Protected participant: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Patient hospitalized without consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2027-05-21 (Estimated); Study Completion 2027-09-21 (Estimated)

PRIMARY OUTCOMES:
Compare the success rate of outpatient treatment of the V-Notes route and the conventional laparoscopic route and to compare the success rate of outpatient treatment of the V-Notes route and the robot-assisted laparoscopic route. | 6 hours post-surgery
  Success rate of outpatient treatment

SECONDARY OUTCOMES:
Compare the success rate he success rate of outpatient treatment of the conventional laparoscopic route and the robot-assisted laparoscopic route. | 6 hours post-surgery
  Success rate of outpatient treatment
Compare the readmission rate in post-operative night for all patients. | 24 hours post-surgery
  Readmission rate
Compare the readmission rate within 7 days post-surgery for all patients. | 7 days post-surgery
  Readmission rate
Evaluate the reason for the failure of outpatient treatment | 6 hours post-surgery
  Rate of failure of outpatient treatment coming from the patient Rate of failure of outpatient treatment coming from the surgeon Rate of failure of outpatient treatment coming from the entourage Rate of failure of outpatient treatment coming from other reason
Compare patient satisfaction for all technique by 5-modal Likert scale | 3 months post-surgery
  Satisfaction assessed by 5-modal Likert scale :
  "Are you satisfied with the outpatient management of benign total hysterectomy? Very dissatisfied/ dissatisfied/ neither satisfied nor dissatisfied/ satisfied/ very satisfied"
Compare patient satisfaction for all techniques by her opinion on: if this had to be done again (yes/no) | 3 months post-surgery
  Satisfaction assessed by the following question :
  If you had to do it again, would you accept outpatient care for this type of surgery? (yes/no)
Compare the occurence of intraoperative adverse events and up to one month postoperatively. | 1 month post-surgery
  Intraoperative and postoperative adverse events related to hysterectomy
Evaluate sequelae for all surgical approaches. | 3 months post-surgery
  Sequelae of the surgical approach
Evaluate post-operative pain by Digital scale. | 6 hours post-surgery
  Digital pain scale (From 0 to 10) before leaving the recovery room (SSPI) and post-operatively before leaving the hospital
Evaluate the use of analgesic. | 8 days post-surgery
  Type of analgesic and number of analgesic tablets actually taken by the patient in the 8 post-operative days.
Compare patient's Hospital Anxiety and Depression Scale score during their treatment. | baseline, 1 month post-surgery, 3 months post-surgery
  HADS (Hospital Anxiety and Depression Scale) is a self questionnaire including 14 items which identifies and quantifies the depression and anxiety from which a person suffers.
  7 questions relate to anxiety (total A) and 7 others to the depressive dimension (total D), allowing thus obtaining two scores (maximum score of each score = 21). A higher score indicates higher distress.
Compare patient's quality of life. | baseline, 1 month post-surgery, 3 months post-surgery
  The patient's quality of life will be measured by EQ-5D-5L. It essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Compare the recuperation of sexual function between baseline and 3 months post-surgery. | baseline, 3 months post-surgery
  PISQ-12 is a validated and reliable short form that evaluates sexual function in women with urinary incontinence and/or pelvic organ prolapse
Compare the resumption of usual activity and work. | 3 months post-surgery
  Resumption of usual activity (duration of incapacity) and professional activity (duration of work stoppage)
Compare intraoperative bleeding. | Day of surgery
  Intraoperative bleeding will be evaluated by suction jar decreased by the amount of washing
Compare hemoglobin decrease during intervention. | Day of surgery
  Difference in hemoglobin between pre-operative and post-operative assessment (if applicable)
Compare skin-to-skin duration. | Day of surgery
  Skin-to-skin duration of the procedure between incision and closure
Compare room occupancy time. | 3 months post-surgery
  Room occupancy time defined between the time of entry and exit of the patient from the operating room
Evaluate the medico-economic value of the use of each technique. | 3 months post-surgery
  Cost-utility ratio of the use of each technique

CONTACTS AND LOCATIONS:
Locations (1):
- Polyclinique Jean Villar, Bruges, France

IPD SHARING:
Plan to Share IPD: No